CLINICAL TRIAL: NCT06729060
Title: Do the Effects of Mental Fatigue on Reaction Time and Game Performance in Esport Players Change With Motor Imagery?
Brief Title: Mental Fatigue on Reaction Time and Game Performance in Esport Players
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Bandırma Onyedi Eylül University (Other)
Collaborators: The Scientific and Technological Research Council of Turkey (Other)
Responsible Party: Principal Investigator, Ozan Bahadır Turkmen, Research Assistant, Bandırma Onyedi Eylül University
Allocation: Randomized | Model: Factorial | Masking: Double | Purpose: Treatment
Other Study IDs: 2024-18-28
Record Dates: First submitted 2024-09-27; First posted 2024-12-11 (Actual); Last update posted 2025-09-16 (Actual); Status verified 2025-03

CONDITIONS: Esport Players; Gaming Performance; Mental Fatigue
Keywords: esport players; mental fatigue; motor imagery
MeSH Terms: conditions — Mental Fatigue | interventions — Physical Functional Performance

STUDY DESIGN:
Intervention Model Description: The study has a randomised controlled single-blind experimental design.
Who Masked: Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (3):
- Control Group (No Intervention)
- Combination of Motor Imagery and Physical Performance Group (Active Comparator): For 15 minutes you will physically eliminate targets by clicking on them in the Aim Lab Trainer (Physical Performance Part).
  Then, on a screen divided into 60 squares, the target will appear and disappear in a random square for 5 seconds. At the same time, the metronome will give a warning sound at each new target. The stimulus will come every five seconds and each time the stimulus comes, the target will imagine that it has disappeared. In the next 5 seconds, the stimulus will come again in a different place and he will imagine that he has destroyed it again. In the first two weeks, this will happen for 60 stimuli with 5 second intervals.
  (60target*5sec=300sec *3=900sec/60 =15 min). In the next 2 weeks, the interval will be reduced by 1 second and in the last two weeks it will not be reduced. But the duration will always be 15 minutes (Motor Imagery Part).
  Interventions: Other: Combination of Motor Imagery and Physical Performance
- Physical Performance Group (Active Comparator): For 30 minutes, they will eliminate the Aim Lab Trainer test by clicking quickly and accurately with their dominant hands. The physical performance application to be applied both in this group and in the Motor Imagery and Physical Performance Combination Group is the same and will be applied in the same way for 8 weeks.
  Interventions: Other: Physical Performance

INTERVENTIONS:
Other: Combination of Motor Imagery and Physical Performance — For 15 minutes you will physically eliminate targets by clicking on them in the Aim Lab Trainer (Physical Performance Part).
  Then, on a screen divided into 60 squares, the target will appear and disappear in a random square for 5 seconds. At the same time, the metronome will give a warning sound at each new target. The stimulus will come every five seconds and each time the stimulus comes, the target will imagine that it has disappeared. In the next 5 seconds, the stimulus will come again in a different place and he will imagine that he has destroyed it again. In the first two weeks, this will happen for 60 stimuli with 5 second intervals.
  (60target*5sec=300sec *3=900sec/60 =15 min). In the next 2 weeks, the interval will be reduced by 1 second and in the last two weeks it will not be reduced. But the duration will always be 15 minutes (Motor Imagery Part).
  Arms: Combination of Motor Imagery and Physical Performance Group
Other: Physical Performance — For 30 minutes, they will eliminate the Aim Lab Trainer test by clicking quickly and accurately with their dominant hands. The physical performance practice to be applied both in this group and in the Motor Imagery and Physical Performance Combination Group is the same and will be applied in the same way for 8 weeks
  Arms: Physical Performance Group

SUMMARY:
Electronic sports (e-sports) gained popularity in the early 2000s within the computer gaming community and reached an audience of approximately 395 million people worldwide by 2018 (Bányai et al., 2019; Nagorsky and Wiemeyer, 2020). The exponential growth of e-sports globally has led to its recognition as a sport, creating employment opportunities for players who master and showcase game-related skills, turning e-sports players into professional athletes supported by well-known companies, and providing the chance to win large cash prizes (Seo, 2013; Giakoni-Ramírez et al., 2022). As a result of this progress, it is estimated that the number of global players could reach 3.38 million in 2023, with revenues reaching $184.0 billion (Report, 2023). E-sports refers to competitive video games where teams or individuals compete against each other, and it is recognized as a sport activity that helps players develop and train their mental skills and hand-eye coordination (Adamus, 2012). Although it requires less physical activity and contact compared to most sports, e-sports shares some common aspects with traditional athletic sports. For instance, in games divided into tournaments and matches, players either individually or as a team face off against opponents. Other commonalities include players often practicing for hours every day, working professionally, and being able to secure sponsorships from companies (Jacobs, 2015). There are various computer games with different mechanics and competition rules that players must master. To reach and maintain peak performance, players need to continually exercise and improve their skills and abilities (Nagorsky and Wiemeyer, 2020). E-sports players must adapt their hand-eye coordination, respond quickly to changing conditions, and continuously adjust their reaction speeds (Steenbergen et al., 2015; Stewart et al., 2020; Urbaniak et al., 2020). Key components of e-sports performance include hitting accuracy for moving targets that quickly appear on the screen (hit accuracy) and rapid response to stimuli (reduced reaction time). In the literature, it has been observed that reaction time and hit accuracy are commonly evaluated to measure an e-sports player's performance (Koposov et al., 2020; Sainz et al., 2020; Luu et al., 2021; Ersin et al., 2022). Nagorsky and colleagues have stated that reaction time is the most important performance indicator in all e-sports disciplines (Nagorsky and Wiemeyer, 2020). Since reduced reaction time is crucial for the quick execution of decisions, it can be a factor that makes a difference in e-sports (Brandmeyer et al., 2021). According to recent literature, the Aim Lab software is one program that can measure and improve e-sports player performance (Roldan and Prasetyo, 2021). Researchers plan to use reaction time, hit accuracy, and the Aim Lab training application to evaluate e-sports players' performance. Mental fatigue is a psychobiological state that arises from prolonged cognitive activities (Marcora et al., 2009). It has been shown in the literature that mental fatigue induced by a protocol (e.g., the commonly used Stroop Test) reduces performance parameters such as running and total distance in various team sports (Smith et al., 2015), impairs running, passing, and shooting performance specific to soccer (Smith et al., 2016), and similarly negatively affects physical performance in cricket (Veness et al., 2017) and Australian football players (Weerakkody et al., 2021). Additionally, it has been reported that mental fatigue induced by the Stroop test affects passing decisions in professional soccer players (Gantois et al., 2020) and decreases decision-making performance in sub-elite soccer players (Trecroci et al., 2020).

Furthermore, it has been shown that playing sports-based video games or using social media also causes mental fatigue, negatively affecting decision-making and visuomotor skills (Fortes et al., 2020; Fortes et al., 2022; Fortes et al., 2023). Although the literature generally indicates that playing video games or using social media leads to mental fatigue, there are also studies suggesting otherwise. Ciocca and colleagues found that a 30-minute video-based tactical task did not cause mental fatigue and did not negatively affect physical or technical performance (Ciocca et al., 2022). For all these reasons, it is important to apply a structured fatigue protocol to ensure that the individual is genuinely mentally fatigued. Therefore, in our study, the 30-minute Stroop test will be used to induce mental fatigue, focusing on this gap in the literature.

ELIGIBILITY:
Inclusion Criteria:

* Being between the ages of 18-30: This age range was chosen because it is the age group with the highest number of e-sports players. After the age of 30, both the number of e-sports players decreases and reaction times decrease with age, so researchers accepted the age of 30 as a cut-off value.
* Male gender: E-sportsmen are generally composed of men. In addition to the difficulty of reaching female e-sportsmen, female e-sportsmen will not be included since it is known that performance parameters evaluated in heterogeneous groups will lead to differences.
* Doing e-sports for at least 6 hours or more per week for at least 6 months.

Exclusion Criteria:

Without Study

* Having any neurological, visual or auditory impairment,
* Having undergone any upper extremity surgery,
* Those who meet the recruitment criteria but are unable to come to the laboratory Those who used any medication or performance-enhancing dietary supplement in the month before the study Exclusion from the Evaluation Day in the Study: Participants will be questioned verbally before the evaluation and participants who do not meet the criteria will not be evaluated that day. After 1 day, they will be re-evaluated.
* Taking medication known to have stimulant or sedative effects
* Consumption of alcohol at least 24 hours before
* Consuming caffeine at least 8 hours before Exclusion from Intervention Groups: Participants who violate these criteria during the intervention will be excluded from the study.
* Those who take part in the intervention groups and are absent 20% or more
* Changes in initial physical activity categories according to the results of the International Physical Activity Scale Short Form

Ages: 18 Years to 30 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Gender Based: Yes
Enrollment: 45 (Actual)
Dates: Start 2024-09-01 (Actual); Primary Completion 2025-04-15 (Actual); Study Completion 2025-06-01 (Actual)

PRIMARY OUTCOMES:
Game Performance-Aim Lab Trainer | 8 weeks
  Aim Lab Trainer Testi Aim Lab is a personal training tool designed to assist players in developing their skills. It offers a range of features, including goal analysis, feedback, and a speed tap, which are intended to enhance the player's core abilities, including perception, movement, and more. At the commencement of the test, the participant will endeavour to rapidly and accurately target the 60 displayed targets on the screen. At the conclusion of the test, the mean time per target of the ms category will be calculated. The test will be repeated three times, and the highest score will be recorded. Following each trial, a three-minute interval will be observed. In order to encourage participants to utilise the mouse in order to "tap" the screen with a single touch, the test will be conducted using the digital distribution platform Steam and the free-to-use Aim Lab application (https://store.steampowered.com/app/714010/Aim_Lab).
Visual Reaction Time Test | 8 weeks
  The participant will be asked to place the index finger of the dominant hand on the left button of a computer mouse and press the left button as soon as the green lights up on the traffic light shape on the screen. The time between the light stimulus and the participant's response will be recorded in milliseconds. The tester will press the 'start' button on the screen to initiate the next trial. The built-in variable delay of 1-5 seconds will eliminate possible cues that may help the participant each time the tester presses the 'start' button. The test will be administered five times and the average will be calculated as the test score (measured in milliseconds) (Lord et al. 2003). The website (https://humanbenchmark.com/tests/reactiontime) will be used for simple reaction time measurement.
Auditory Reaction Time Test | 8 weeks
  Participants will be asked to click on the 'space' key every time they hear a sound. After five applications, data will be taken from the out
Fatigue Assessment | 8 weeks
  Perceived fatigue severity will be assessed with the Borg scale, which is widely used in the assessment of fatigue severity. The level of mental fatigue felt by the participants is scored between 0 and 10 and an increase in the value indicates an increase in the severity of fatigue (Borg 1982). This scale will be used to determine the general level of mental fatigue perceived by the participants at the beginning of the assessment day before the tests started and at the end of the day after all the tests.

SECONDARY OUTCOMES:
International Physical Activity Questionnaire-Short Form | 8 weeks
  Physical activity level will be evaluated with the International Physical Activity Questionnaire (Short Form). International validity and reliability study of the questionnaire was conducted by Craig et al. (Craig et al., 2003) and Turkish validity and reliability study was conducted by Saglam et al. (Saglam et al., 2010). The questions in the questionnaire were developed to be used by adults aged 18-65 years. The questionnaire assesses the time spent on vigorous and moderate physical activity, walking and sitting in the last 7 days. The time spent sitting is not included in the scoring of the test, but is expressed as a separate indicator (Craig et al., 2003). Scoring is calculated by multiplying the MET level of the activity (multiples of resting oxygen consumption), the number of days per week and the number of minutes per day. Severe physical activity is 8 METs, moderate physical activity is 4 METs, walking is 3.3 METs and sitting is 1 MET (Craig et al., 2003; Orhan et al. 2015;

CONTACTS AND LOCATIONS:
Locations (1):
- Bandırma Onyedi Eylül University Physical Therapy and Rehabilitation, Bandırma, Balıkesir, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No